CLINICAL TRIAL: NCT04805086
Title: Phase I/II MONACO Cell Therapy Study: Monocytes as an Anti-fibrotic Treatment After COVID-19
Brief Title: The MONACO Cell Therapy Study: Monocytes as an Anti-fibrotic Treatment After COVID-19
Acronym: MONACO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 289624
Record Dates: First submitted 2021-03-03; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Fibrosis; Interstitial Lung Disease; Covid19
Keywords: Phase I/II; cell therapy; ATIMP
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; COVID-19 | interventions — MON002

STUDY DESIGN:
Intervention Model Description: Prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MON002 (Experimental): Minimum of 1x10~7 cells to maximum of 2x10~6 cells/kg. Single infusion.
  Interventions: Biological: MON002

INTERVENTIONS:
Biological: MON002 — Autologous monocytes

SUMMARY:
Up to a third of patients who recovered from SARS coronavirus (SARS-CoV) had a 20% decline in lung function with a long term reduction in exercise capacity and SF-36 health status a year after infection. Similar outcomes are now being reported in COVID-19 patients, with interstitial lung disease (fibrosis) and long term lung function decline being a common feature. Anti-fibrotic monocytes/macrophages are important for the clearance of partially degraded collagen fragments of fibrotic extracellular matrix, in particular fibrillary-type collagen.

MON002 is an autologous monocyte product, cultured in vitro prior to intravenous delivery into patients with post-COVID-19 lung fibrosis.

DETAILED DESCRIPTION:
The MONACO Cell Therapy Study is a prospective, non-randomised, open label study phase I/II clinical trial with a key objective of evaluating safety of MON002 in 5 adults who have a clinical diagnosis of interstitial lung disease (pulmonary fibrosis) after recovery from acute COVID-19 infection. The main objectives of this study are to: (1) to determine the safety profile of MON002 by assessing clinical responses in adults with post-COVID-19 pulmonary fibrosis and (2) to assess its impact on reducing disease morbidity/severity in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical evidence/diagnosis of interstitial lung disease (fibrosis) following COVID-19 infection
2. Aged at least 18 years
3. Willing and able to participate in the MONACO Cell Therapy Study
4. Signed and dated written informed consent.

Exclusion Criteria:

1. Subjects who have had other investigational medicinal products within 90 days prior to screening or during the treatment phase.
2. Malignant or premalignant haematological conditions
3. Serologically positive for antiHIV1,2; HBsAg; Anti-HBc; Anti-HCVab;Anti-HTLV1,2 or syphilis (Treponema palladium)
4. Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully treated non metastatic basal/squamous cell carcinoma of the skin)
5. Evidence of significant local or systemic infection
6. Any uncontrolled medical condition or concurrent disease that could interfere with the study objectives
7. Clinical diagnosis of interstitial lung disease prior to the COVID-19 infection
8. Any condition which, in the judgement of the Investigator, would place the subject at undue risk
9. Female patients of childbearing potential with a positive serum pregnancy test at enrolment
10. Sexually active Women of Childbearing Potential who do not agree continued abstinence from heterosexual intercourse or to use highly effective methods of birth control for the duration up to 4 weeks post IMP administration. Men who do not agree to use a condom if their partner is of child bearing potential, even if they have had a successful vasectomy after receiving the therapy
11. Female patients who are breastfeeding
12. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow up visit schedule
13. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
14. Patients unable to freely give their informed consent (e.g. individuals under legal guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-03-08 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of serious adverse events (SAE) related to the administration of the IMP | Total number of SAEs at 12 months after administration
  Any SAEs that result in death, are life-threatening, require hospitalisation or prolonged or existing hospitalisation (that are not determined to be as a result of disease progression) or result in persistent or significant disability or incapacity

SECONDARY OUTCOMES:
Absolute change from baseline of predicted forced vital capacity (FVC) | 3, 6 and 12 months
Rate of decrease in FVC | 3, 6 and 12 months
Time to first occurrence of a ≥10% absolute decline in percentage of predicted FVC | 3, 6 and 12 months
Time to decrease from baseline (relative change) of ≥ 10% in FVC (mL/year) | 3, 6 and 12 months
Time from cell administration to first event of acute pulmonary fibrosis exacerbation | 3, 6 and 12 months
  Defined by (a) worsening or development of dyspnoea and radiologic evidence of new bilateral ground-glass abnormality or consolidation superimposed on a reticular or honeycomb background pattern
Absolute change in transfer capacity of the lung (TLCO). | 3, 6 and 12 months
Improvement in quality of life as indicated by the King's Brief Interstitial Lung Disease (K-BILD) score | 3, 6 and 12 months
  Score is transformed to range from 0-100. 100=best health status
Improvement in quality of life as indicated by the 36-Item Short Form Survey (SF-36) score | 3, 6 and 12 months
  Score is transformed to range from 0-100. 100=best health status
Reduction in fibrosis score on high resolution lung CT | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Patel, PhD FRCS, Study Chair — King's College London and Guy's & St Thomas' NHS Foundation Trust; Bijan Modarai, PhD FRCS, Principal Investigator — King's College London and Guy's & St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided